CLINICAL TRIAL: NCT00342524
Title: Collection of Convalescent SARS Plasma by Apheresis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905192; 05-I-N192
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-02-08

CONDITIONS: Severe Acute Respiratory Syndrome; SARS
Keywords: IVIG; Plasmapheresis; Blood Collection; Immune Globulin; Severe Acute Respiratory Syndrome; SARS
MeSH Terms: conditions — Severe Acute Respiratory Syndrome

SUMMARY:
The purpose of this study is to collect plasma by apheresis from patients who have recovered from Severe Acute Respiratory Syndrome (SARS). This plasma will be processed into a SARS-antibody enriched intravenous immune globulin (IVIG) product. This product will then be available for use in a clinical trial if a SARS epidemic recurs.

Potentially eligible participants are people between 18 and 56 years of age who have recovered from SARS. Potential participants will undergo three sequential screenings to determine their eligibility for this study. Eligible participants will then be scheduled for plasmapheresis. After apheresis, additional testing will be performed on a sample of the source plasma. Once the sample has been tested and cleared, the source plasma will be shipped to the United States to the storage facility and finally to the site of manufacturing of the IVIG product. Participants may donate plasma again after 14 days.

The study will not have a direct benefit for participants. However, participation may help develop a treatment that could be useful to other people who become infected with SARS.

DETAILED DESCRIPTION:
Beginning in February 2003, there was an outbreak with a novel coronavirus causing an atypical pneumonia, subsequently referred to as Severe Acute Respiratory Syndrome (SARS). This syndrome is associated with a high mortality rate and has no proven treatment. There is, however, some evidence that treatment with convalescent plasma was beneficial.

The primary purpose of this protocol is to collect plasma by apheresis from patients that recovered from SARS, and process this plasma into a high titer anti-SARS intravenous immune globulin (IVIG). This will be a collaboration between the National Institute of Allergy and Infectious Diseases and the Chinese University of Hong Kong. Cangene Corporation has been contracted to manufacture the collected plasma in the United States (U.S.) into an IVIG product, which can then be used for pre-clinical efficacy studies under an IND in a clinical trial if SARS recurs. It is intended that the treatment trial would be conducted in Hong Kong and/or the U.S., as well as any other place the disease recurs.

ELIGIBILITY:
* INCLUSION CRITERIA:

RECOVERED SARS SCREENING - INCLUSION CRITERIA (ALL OF THE FOLLOWING):

1. Clinical diagnosis of SARS occurring greater than or equal to 3 months prior to screening. (objective documentation of SARS is not necessary)
2. The ability to understand and willingness to sign a written consent form and comply with study requirements and procedures.

SARS APHERESIS SCREENING - INCLUSION CRITERIA (ALL OF THE FOLLOWING):

1. SARS Ab level greater than or equal to 1:80
2. Adequate clinical parameters (must meet all of the criteria below):

   1. Afebrile (temperature less than 38 degrees C)
   2. Systolic blood pressure greater than 100 and less than 160 mmHg
   3. Diastolic blood pressure greater than 50 and less than 100 mmHg
   4. Heart rate between 50-100 beats/minute
   5. Weight greater than or equal to 110 pounds (50kg)
3. Adequate laboratory parameters (must meet all of the criteria below):

   1. Hemoglobin greater than or equal to 12.5 g/dL for females or 13 grams/dL for males
   2. HCT greater than or equal to 38%
   3. Platelets greater than or equal to 150,000 x 10(3)/microL
   4. Total serum protein greater than or equal to 6.0 grams/100 milliliters of blood
   5. ALT less than 1.5 Upper limit of normal
   6. Quantitative immune globulin levels (all of the following):

      * Ig A greater than or equal to 90 mg/dL
      * Ig G greater than or equal to 650 mg/dL
      * Ig M greater than or equal to 35 mg/dL
4. Negative tests for blood borne pathogens (must meet all of the criteria below):

   1. Human Immunodeficiency Virus 1/2 Antibody (Anti-HIV1/2) negative
   2. Hepatitis B virus surface antigen (HBsAg) negative
   3. Hepatitis C virus antibody (anti-HCV) negative
   4. RPR non-reactive
   5. HTLV antibody
5. Adequate peripheral venous access for plasmapheresis (as judged by the examiner)

DAY OF DONATION SCREENING - INCLUSION CRITERIA:

1. Afebrile (temperature less than 38 degrees C)
2. Systolic blood pressure greater than 100 and less than 160 mmHg
3. Diastolic blood pressure greater than 50 and less than 100 mmHg
4. Heart rate between 50-100 beats/minute
5. Blood hemoglobin level of greater than or equal to 12.5 grams/dL for females or 13 grams/dL for males
6. Total serum protein greater than or equal to 6.0 grams/100 milliliters of blood
7. Weight greater than or equal to 110 pounds (50kg)
8. RPR performed in the 4 months prior to the day of donation and non-reactive.
9. AST performed in the 4 months prior to the day of donation less than 1.5 upper limit of normal.
10. SARS antibody performed in the 4 months prior to the day of donation, and Ab titer greater than or equal to 1:80
11. Quantitative immune globulin levels performed in the 4 months prior to the day of donation (and all of the following):

    * Ig A greater than or equal to 90 mg/dL
    * Ig G greater than or equal to 650 mg/dL
    * Ig M greater than or equal to 35 mg/dL

EXCLUSION CRITERIA:

RECOVERED SARS SCREENING - EXCLUSION CRITERIA:

1. Age less than 18 years old, or greater than 56 years old.
2. Signs of active respiratory infection including cough, dyspnea, or oxygen requirement.
3. Subjective fever in the last 3 days
4. History of headache with fever within the past 7 days.
5. Known history of congestive heart failure, pulmonary hypertension or other diseases in which the fluid shifts associated with apheresis present more than minimal risk.
6. Known history of bleeding diathesis or therapeutic anticoagulation.
7. Bilateral mastectomy or other relative contraindications to peripheral venous catheter insertion.
8. Within the last week has:

   * Taken traditional Chinese medicines.
   * Received hepatitis B vaccination.
9. Within the last 3 weeks has:

   - Received live-attenuated vaccines such as BCG, yellow fever, measles, mumps, poliomyelitis (oral), or live attenuated typhoid fever.
10. Within the last 4 weeks has:

    - Received rubella or varicella zoster (chicken pox) vaccination.
11. Within the last 6 weeks has:

    * Received standard IVIG for hepatitis A or other indications.
    * Received anti-tetanus toxoid or other passive immunizations with animal serum.
    * Been diagnosed with West Nile virus infection.
12. Within the last 8 weeks:

    - Was vaccinated with the small pox vaccine, or was in close contact with someone who was vaccinated (i.e., close family member).
13. Within the last 3 months has:

    * A history of unexplained weight loss of more than 10 lbs/4.5 kg.
    * Has been seen by a physician or public health staff for investigation of TB.
    * Current or previous participation in any other apheresis procedures/protocols (not related to this protocol).
14. Within the last 6 months has had:

    * A diagnosis of Dengue fever.
    * An induced abortion.
    * A blood donation of a double unit of red cells.
15. Within the last 12 months has:

    * Received any blood or blood component.
    * Donated blood at a paid donation center (donations at a hospital blood bank do not apply).
    * History of unsafe (multiple-use equipment) tattoo, acupuncture, or piercing practices.
    * Received an organ transplant.
    * Received a bone or skin graft.
    * Lived with someone who has any type of hepatitis.
    * Traveled to areas with malaria.
    * Incarcerated for more than 72 hours.
    * Oral or inhalation use of illegal drugs (i.e. those not prescribed by a physician).
    * Received hepatitis B IVIG for passive immunity.
16. Within the last 12 months has had sexual contact with (any of the following):

    * An individual having viral hepatitis.
    * A prostitute or anyone else who takes money or drugs or other payment for sex.
    * Anyone who has ever used needles to take drugs, steroids, or anything else not prescribed by their doctor.
    * Anyone who has hemophilia or has used clotting factor concentrates.
    * For females, a male who has ever had sexual contact with another male.
17. Within the last 2 years has:

    - Has received treatment for tuberculosis.
18. Within the last 3 years:

    - Has been diagnosed with malaria.
19. History of cancer that meets any one of the following criteria:

    * Non-melanoma skin cancers within the last 1 year
    * Melanoma or any other cancer (excluding non-melanoma skin cancers).
20. Medication history that includes any of the following:

    * Finasteride (Proscar, Propecia) within the last 1 month.
    * Isotretinoin (Accutane) within the last 1 month.
    * Acitretin (Soriatane) within the last 3 years.
    * Etretinate (Tegison) at any time.
    * Dutasteride (Avodart) within the last 6 months.
    * Viagra within the last week.
    * Growth hormone made from human pituitary glands at any time
    * Any growth hormone administered prior to 1985.
    * Beef insulin from the United Kingdom at any time.
    * Xenical or other weight reduction medications within the last week.
21. Has ever had (any of the following)

    * Known history of HIV.
    * Sexual contact with someone known to have HIV or HTLV.
    * Known history of Hepatitis after the 11th birthday.
    * Had a relative with Creutzfield-Jakob Disease, or been told that this disease is inherited within the family.
    * Received blood transfusion in the United Kingdom.
    * History of receiving money, drugs or other payment for sex.
    * History of receiving clotting factor concentrates.
    * History of a dura mater graft.
    * History of babesiosis.
    * For male donors, history of sexual contact with another male.
    * Used needles to take drugs, steroids, or other medications not prescribed by a physician.
    * Trypanosomiasis (Chagas' disease and sleeping sickness)
    * Leshmaniasis (Kala-azar)
    * Filariasis
    * Q fever
    * Yaws
    * All venereal diseases (including genital herpes)
    * Sexual contact with anyone who lived in listed African countries after 1977.
22. History of living 3 or more months in the UK from 1980-1996.
23. History of living 5 or more years in Europe since 1980.
24. Currently pregnant (if known).

SARS APHERESIS SCREENING - EXCLUSION CRITERIA:

1. Positive urine pregnancy test.

DAY OF DONATION SCREENING - EXCLUSION CRITERIA:

1. Blood hemoglobin greater than or equal to 17 for males or females.
2. Pilots, fireman, scaffolding workers, divers, bus and truck drivers, crane operators or underground workers who are on duty or planned to work the day of donation.
3. Planned participation in dangerous sports such as rock climbing, hang gliding, or scuba-diving the day of donation.
4. Signs/symptoms of an acute respiratory disease.
5. Signs/symptoms of any skin disease at the site of phlebotomy or any such disease generalized to such an extent as to create a risk of contamination of the plasma.
6. Skin punctures or scars indicative of addiction to self-injected narcotics.
7. Persons with signs of debilitation, under nutrition, plethora, anaemia, jaundice, cyanosis, dyspnea, or mental instability.\
8. In the opinion of the interviewer, a donor that: (either of the following)

   * appears to be under the influence of any drug or alcohol
   * for any reason does not appear to be providing reliable answers to medical history questions
9. Within the last 8 weeks, has not had the red blood cells returned during a plasmapheresis procedure.
10. Within the last 8 weeks has been a donor of a unit of whole blood.
11. Subjective fever or other symptoms suggestive of active infection.
12. Known exposure (since screening or previous donation) to HIV, Hepatitis B or Hepatitis C.
13. Received toxoid, killed vaccines, or recombinant vaccines such as cholera, typhoid, diphtheria, tetanus, hepatitis A, influenza, poliomyelitis (injection), or pertussis within the last 24 hours.
14. Received live-attenuated vaccines such as BCG, yellow fever, measles, mumps, poliomyelitis (oral), or live attenuated typhoid fever within the last 3 weeks.
15. Received rubella or varicella zoster (chicken pox) vaccination within the last 4 weeks.
16. Current or previous participation (within the last 3 months) in any other apheresis procedures/protocols (i.e. not related to this protocol).
17. Known or suspected pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-07-06; Study Completion 2007-02-08

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Background] Fouchier RA, Kuiken T, Schutten M, van Amerongen G, van Doornum GJ, van den Hoogen BG, Peiris M, Lim W, Stohr K, Osterhaus AD. Aetiology: Koch's postulates fulfilled for SARS virus. Nature. 2003 May 15;423(6937):240. doi: 10.1038/423240a. PMID 12748632